CLINICAL TRIAL: NCT05133414
Title: Effects of Selective Left Subclavian Ansae Stimulation on Human Cardiac Electrophysiological Properties - a Potential Percutaneous Target for Neuromodulation in Atrial Fibrillation.
Brief Title: Subclavian Ansae Stimulation in AF (SAS-AF)
Acronym: (SAS-AF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 303347
Record Dates: First submitted 2021-11-01; First posted 2021-11-24 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Subclavian ansae stimulation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants will receive stimulation of the left subclavian ansae. (Experimental): Participants as self-controlled cases for the study. Human cardiac haemodynamics and electrophysiological in response to left subclavian ansae stimulation will be studied.
  Interventions: Other: Selective left subclavian ansae stimulation

INTERVENTIONS:
Other: Selective left subclavian ansae stimulation — Percutaneous, transarterial approach for target stimulation

SUMMARY:
Atrial Fibrillation (AF) is a common heart rhythm condition that affects over 3% of the total population. AF can lead to serious health problems such as heart failure or stroke and can also cause troublesome symptoms in some people. Although many advances have been made, there remains a pressing need to improvement treatment of AF.

It is increasingly recognised that the brain and nerves can influence the electrical activity of the heart.

Therefore, this research involves studying a new nerve target (Subclavian ansae) that is connected to the heart and can be a potential target for future treatment of AF. This nerve lies around an area close to an artery that runs to participant's left arm called left subclavian artery which can be approached via leg (key hole). The investigators aim to conduct this study in patients who have been referred for first time AF ablation.

DETAILED DESCRIPTION:
Atrial Fibrillation (AF) is a common and significant medical problem that affects approximately 3% of the population. There is increasing recognition of the importance of interactions between the heart and the autonomic nervous system (ANS) in the pathophysiology of arrhythmias. The role of ANS in the onset and maintenance of AF is thought to be related to autonomic imbalance. Several studies have experimented the use of autonomic modification in AF and identified potential targets for therapy ( for example: ganglionic plexi ablation, renal denervation, stellate ganglion block, and low level vagal nerve stimulation). However, some targets like stellate ganglion block/sympathectomy will have off-target side-effects. Easily accessible, minimally invasive, and selective targets for neuromodulation are of great interest for development of novel therapy in the management of AF.

The subclavian ansae was first described in 1864 by Vieussens and is a nerve cord that forms a loop inferiorly around the subclavian artery and connects the inferior cervical ganglion and middle cervical ganglia.According to literature cardiac-related preganglionic fibers arising from the thoracic cord traverse up the paravertebral chain through the T1-T2 region, some making synaptic contact with postganglionic neurons in the stellate with others projecting through the subclavian ansae to more distal intrathoracic ganglia (middle cervical, mediastinal, and intrinsic). As such the ansa subclavia and the T1-T2 region of the paravertebral chain are critical nexus points for sympathetic nerve traffic to and afferent projections of the heart. Based on structure and function consideration, both sites are potential targets for cardiac neuromodulation.

Preclinical studies have showed that stimulation of the subclavian ansae produces reproducible increases in cardiac rate, contractility and conduction velocity. Denervation of the subclavian ansae followed by stellate ganglion stimulation results in no change in cardiac indices confirming the nodal intervention point for cardiac sympathetic traffic. Due to the close anatomical proximity, stimulation of subclavian ansae should be possible via the subclavian artery which is accessible by percutaneous approach.

Hypothesis:

The investigators intend to introduce a percutaneous approach for identification and stimulation of subclavian ansae (sympathetic nerves) which exclusively innervate the heart and therefore stimulation will result in in changes in human cardiac haemodynamic and electrophysiological parameters.

Primary objective:

The primary objective of the study is to determine the human cardiac haemodynamics and electrophysiological response to left subclavian ansae stimulation (SAS) in patients with AF.

Secondary objective:

To determine appropriate stimulation parameters to selectively target subclavian ansae via percutaneous transarterial approach and to confirm safety of the procedure.

Patients referred by Electrophysiologist for catheter ablation of paroxysmal AF (PAF) will be recruited. Participants will undergo consenting for the procedure and their involvement in the research study. The procedure will be performed under general anaesthesia. A stimulation wire will be passed into the left subclavian artery via the femoral arterial access. Further wires will be passed (via venous access) to the left top chamber of the heart which will then be used for 3D guided AF ablation after stimulation protocol. Study measurements will be gathered before and after the stimulation subclavian ansae. This will be followed by AF ablation (pulmonary vein isolation) and direct current cardioversion (DCCV) [if required] as standard care.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Age 18-80 years
* First time PAF ablation

Exclusion Criteria:

* Creatinine clearance (eGFR) < 30mls/min
* Contraindication or unable to take anticoagulation
* Uncontrolled hypertension
* Contraindication for catheter ablation
* BMI > 35
* Haemodynamically unstable
* Recent Stroke/ myocardial infarction
* Significant carotid artery stenosis
* Significant carotid artery stenosis or peripheral arterial disease
* Allergy to contrast
* Presence of pacemaker or implantable cardioverter defibrillator (ICD)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Measuring the rate of change in heart rate (beats per minute) in response to subclavian ansae stimulation (SAS). | During index procedure for catheter ablation
  Measuring the change in heart rate during and post stimulation of the SAS compared to baseline measurement at rest through the mapping catheter and surface ECG electrodes.
Measuring the rate of change in blood pressure (mmHg) in response to subclavian ansae stimulation (SAS). | During index procedure for catheter ablation
  Measuring the blood pressure (systolic and diastolic) through the arterial line during and post stimulation of the SAS compared to baseline measurements at rest.
Measuring the rate of change in conduction velocity (m/s) within left and right atrium in response to subclavian ansae stimulation (SAS). | During index procedure for catheter ablation
  Measuring the conduction velocity in each atrium and changes between the atrial conduction using the intra cardiac catheter electrodes post SAS stimulation comparing with baseline measurements at rest.
Measuring the rate of change in action potential duration (ms) and effective refractive period (ms) in response to subclavian ansae stimulation (SAS). | During index procedure for catheter ablation
  Measurements taken in both atria using the intra cardiac catheter electrodes post SAS stimulation compared to baseline measurements at rest.
Proportion of participants where AF is inducible in response to Subclavian ansae stimulation | During index procedure for catheter ablation
  Number of participants where AF is inducible in response to selective left subclavian ansae stimulation.

SECONDARY OUTCOMES:
Determining the optimal output threshold (Volts/Kg) to selectively stimulate left subclavian ansae via the subclavian artery | During index procedure for catheter ablation
  To determine the delivery energy to stimulate the subclavian ansae to achieve 10-20% increase in heart rate from baseline with stimulation in each participants.
Safety and procedure specific complications | During index procedure for catheter ablation
  To assess procedure specific complications related to subclavian ansae stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Finlay, Principal Investigator — Barts Heart Centre
Locations (1):
- Barts Heart Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The data will be anonymous